CLINICAL TRIAL: NCT06664619
Title: A 4-Week, Double-Blind, Placebo-Controlled, Parallel-Group, Efficacy and Safety Trial of Fluticasone Propionate/Albuterol Sulfate Combination Compared to Fluticasone Propionate, Albuterol Sulfate or Placebo Delivered by Multidose Dry Powder Inhaler in Participants 12 Years and Older With Asthma
Brief Title: A Randomized, Double-Blind, Placebo-Controlled Trial on Efficacy and Safety of Fluticasone Propionate/Albuterol Sulfate Combination in Participants 12 Years and Older With Asthma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FpA-AS-30093; 2024-517991-39-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Fp/ABS eMDPI (Experimental): Fluticasone propionate/albuterol sulfate multidose dry powder inhaler with electronic module
  Interventions: Drug: Fp/ABS
- Fp eMDPI (Active Comparator): Fluticasone propionate (Fp) dry powder inhaler with an integrated electronic module (eMDPI)
  Interventions: Drug: FP
- ABS eMDPI (Active Comparator): Albuterol sulfate (ABS) dry powder inhaler with an integrated electronic module (eMDPI)
  Interventions: Drug: ABS
- Placebo eMDPI (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fp/ABS — Inhalation powder
  Other Names: fluticasone propionate/albuterol sulfate combination
  Arms: Fp/ABS eMDPI
Drug: FP — Inhalation powder
  Other Names: fluticasone propionate
  Arms: Fp eMDPI
Drug: ABS — Inhalation powder
  Other Names: albuterol sulfate
  Arms: ABS eMDPI
Drug: Placebo — Inhalation powder
  Arms: Placebo eMDPI

SUMMARY:
The primary objective of the trial is to evaluate the efficacy of fluticasone propionate/albuterol sulfate multidose dry powder inhaler with electronic module (Fp/ABS eMDPI).

Secondary objectives are:

* To evaluate the efficacy of Fp/ABS eMDPI administered four times daily
* To evaluate the safety and tolerability of Fp/ABS eMDPI administered four times daily over four weeks
* To investigate the pharmacokinetics of Fp/ABS eMDPI, ABS eMDPI and Fp eMDPI after administration of a single dose

The planned study duration for each participant is approximately 10 weeks, excluding an optional prescreening visit.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a diagnosis of asthma of at least 6 months duration.
* Participants currently receive a beta-agonist (eg, salbutamol [albuterol] or ICS albuterol or ICS-formoterol) as rescue medication with or without asthma controller medication.
* If female, a participant is currently not pregnant, breastfeeding, or attempting to become pregnant (for at least 30 days before the screening visit and throughout the duration of the trial), or is of non-childbearing potential.

NOTE- Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* The participant has a history of life-threatening asthma defined as any history of significant asthma episode(s) requiring intubation, associated with hypercapnia, respiratory arrest, hypoxic seizures or an asthma related syncopal episode.
* The participant has had an upper or lower respiratory tract infection within 2 weeks or has had a confirmed case of COVID-19 within 6 weeks prior to Visit 1. Symptoms of the infection(s) must be completely resolved prior to entering screening.
* The participant is a current smoker and/or has a history of ≥10 pack years history of smoking. A current smoker is defined as any participant who has used any form of tobacco product (including oral) within the past 6 months, or any orally inhaled products including but not limited to cigarettes, beedis, vaping/ e-cigarettes, hookah/waterpipes, or marijuana. Note: participants with a positive urinary cotinine test will be excluded.
* The participant has another confounding underlying lung disorder (eg, chronic obstructive pulmonary disease (COPD), chronic bronchitis, emphysema, bronchiectasis with the need of treatment, cystic fibrosis, pulmonary fibrosis), or participants with a diagnosis of asthma COPD overlap syndrome.

NOTE- Additional criteria apply, please contact the investigator for more information

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 724 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline forced expiratory volume in one second (FEV1) area under the effect curve over 4 weeks | Baseline, Week 4
  Baseline values are averaged on day 1 to get a single value. Area under the effect curve will be calculated using measurements collected between zero and 6 hours after dosing. Baseline-adjusted post-dose FEV1 AUEC0-6h for visits on Day 1 and at Week 4 will be calculated using the trapezoidal rule.
Change from Baseline trough FEV1 at week 4 | Baseline, Week 4

SECONDARY OUTCOMES:
Time to 15% improvement from baseline FEV1 post-dose on day 1 | Baseline to Post-dose on Day 1
Time to 12% improvement from baseline FEV1 post-dose on day 1 | Baseline to Post-dose on Day 1
Duration of 15% increase in FEV1 from baseline post-dose on day 1 | Baseline Pre-dose to Post-dose on Day 1
Asthma Control Questionnaire-6 (ACQ-6) response at week 4 defined as achieving a decrease in score from baseline value of at least 0.5 for participants with a baseline ACQ-6 score of ≥1.5 | Baseline, Week 4
  The ACQ-6 is a validated 6-item asthma assessment tool that has been widely used. Six questions are self-assessments (completed by the participant), 5 questions assessing asthma symptoms: night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing, and 1 question for short-acting bronchodilator use. Each item on the ACQ has a possible score ranging from 0 (no impairment) to 6 (maximum impairment), and the total score is the mean of all responses. The total score ranging from 0 (totally controlled) to 6 (severely uncontrolled) with higher scores indicating maximum impairment.
Asthma Control Test (ACT) score response at week 4 defined as achieving an increase in score from baseline value of at least 3 | Baseline, Week 4
  The Asthma Control Test (ACT) is a participant self-administered tool for identifying those with poorly controlled asthma comprising 5 items, with 4-week recall (on symptoms and daily functioning). It assesses the frequency of shortness of breath and general asthma symptoms, the use of rescue medications, the effect of asthma on daily functioning, and the overall self-assessment of asthma control measured on a 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled). Total scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
Number of participants with at least one treatment-emergent adverse event | Up to Week 4
Number of participants with at least one treatment-emergent serious adverse event | Up to Week 4
Number of participants who withdraw from treatment due to an adverse event | Up to Week 4
Plasma concentration of Fp | Baseline, Week 4
Plasma concentration of ABS | Baseline, Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (133):
- United States (76):
  - Teva Investigational Site 12087, Phoenix, Arizona
  - Teva Investigational Site 12144, Phoenix, Arizona
  - Teva Investigational Site 12104, Tucson, Arizona
  - Teva Investigational Site 12146, Tucson, Arizona
  - Teva Investigational Site 12102, Little Rock, Arkansas
  - Teva Investigational Site 12154, Encinitas, California
  - Teva Investigational Site 12103, Huntington Beach, California
  - Teva Investigational Site 12068, La Palma, California
  - Teva Investigational Site 12152, Laguna Niguel, California
  - Teva Investigational Site 12145, Long Beach, California
  - Teva Investigational Site 12088, Los Angeles, California
  - Teva Investigational Site 12094, Los Angeles, California
  - Teva Investigational Site 12161, Northridge, California
  - Teva Investigational Site 12105, Oxnard, California
  - Teva Investigational Site 12101, Sacramento, California
  - Teva Investigational Site 12064, San Jose, California
  - Teva Investigational Site 12109, Upland, California
  - Teva Investigational Site 12070, Vista, California
  - Teva Investigational Site 12091, Walnut Creek, California
  - Teva Investigational Site 12142, Lakewood, Colorado
  - Teva Investigational Site 12098, Lake City, Florida
  - Teva Investigational Site 12118, Lake Worth, Florida
  - Teva Investigational Site 12079, Melbourne, Florida
  - Teva Investigational Site 12071, Miami, Florida
  - Teva Investigational Site 12074, Miami, Florida
  - Teva Investigational Site 12086, Miami, Florida
  - Teva Investigational Site 12061, Miami, Florida
  - Teva Investigational Site 12097, Miami, Florida
  - Teva Investigational Site 12092, Miami Lakes, Florida
  - Teva Investigational Site 12076, North Miami Beach, Florida
  - Teva Investigational Site 12095, Palmetto Bay, Florida
  - Teva Investigational Site 12075, Pompano Beach, Florida
  - Teva Investigational Site 12078, Tampa, Florida
  - Teva Investigational Site 12156, Boise, Idaho
  - Teva Investigational Site 12162, Westchester, Illinois
  - Teva Investigational Site 12081, Nottingham, Maryland
  - Teva Investigational Site 12106, Towson, Maryland
  - Teva Investigational Site 12157, White Marsh, Maryland
  - Teva Investigational Site 12119, Boston, Massachusetts
  - Teva Investigational Site 12073, Minneapolis, Minnesota
  - Teva Investigational Site 12066, Richfield, Minnesota
  - Teva Investigational Site 12149, Columbia, Missouri
  - Teva Investigational Site 12108, St Louis, Missouri
  - Teva Investigational Site 12089, St Louis, Missouri
  - Teva Investigational Site 12158, Hastings, Nebraska
  - Teva Investigational Site 12160, Las Vegas, Nevada
  - Teva Investigational Site 12150, Las Vegas, Nevada
  - Teva Investigational Site 12110, Jersey City, New Jersey
  - Teva Investigational Site 12115, Charlotte, North Carolina
  - Teva Investigational Site 12085, Raleigh, North Carolina
  - Teva Investigational Site 12063, Toledo, Ohio
  - Teva Investigational Site 12155, Tulsa, Oklahoma
  - Teva Investigational Site 12117, Clackamas, Oregon
  - Teva Investigational Site 12151, Portland, Oregon
  - Teva Investigational Site 12147, Horsham, Pennsylvania
  - Teva Investigational Site 12072, Philadelphia, Pennsylvania
  - Teva Investigational Site 12114, Pittsburgh, Pennsylvania
  - Teva Investigational Site 12067, Columbia, South Carolina
  - Teva Investigational Site 12111, Myrtle Beach, South Carolina
  - Teva Investigational Site 12112, North Charleston, South Carolina
  - Teva Investigational Site 12107, Rock Hill, South Carolina
  - Teva Investigational Site 12083, Austin, Texas
  - Teva Investigational Site 12060, Austin, Texas
  - Teva Investigational Site 12077, Corsicana, Texas
  - Teva Investigational Site 12159, Dallas, Texas
  - Teva Investigational Site 12090, Dallas, Texas
  - Teva Investigational Site 12143, El Paso, Texas
  - Teva Investigational Site 12080, Kingwood, Texas
  - Teva Investigational Site 12096, McKinney, Texas
  - Teva Investigational Site 12113, Mesquite, Texas
  - Teva Investigational Site 12084, Victoria, Texas
  - Teva Investigational Site 12148, Pleasant View, Utah
  - Teva Investigational Site 12082, Salt Lake City, Utah
  - Teva Investigational Site 12153, South Ogden, Utah
  - Teva Investigational Site 12093, Portsmouth, Virginia
  - Teva Investigational Site 12062, Greenfield, Wisconsin
- Argentina (11):
  - Teva Investigational Site 20154, Buenos Aires
  - Teva Investigational Site 20156, Buenos Aires
  - Teva Investigational Site 20150, Córdoba
  - Teva Investigational Site 20145, Mar del Plata
  - Teva Investigational Site 20151, Mar del Plata
  - Teva Investigational Site 20146, Quilmes
  - Teva Investigational Site 20148, Rosario
  - Teva Investigational Site 20155, Rosario
  - Teva Investigational Site 20147, San Juan Bautista
  - Teva Investigational Site 20152, San Miguel de Tucumán
  - Teva Investigational Site 20149, San Miguel de Tucumán
- Bulgaria (11):
  - Teva Investigational Site 59248, Haskovo
  - Teva Investigational Site 59251, Lovech
  - Teva Investigational Site 59249, Montana
  - Teva Investigational Site 59247, Pleven
  - Teva Investigational Site 59256, Sliven
  - Teva Investigational Site 59246, Sofia
  - Teva Investigational Site 59252, Sofia
  - Teva Investigational Site 59253, Sofia
  - Teva Investigational Site 59245, Stara Zagora
  - Teva Investigational Site 59254, Veliko Tarnovo
  - Teva Investigational Site 59250, Vratsa
- Czechia (3):
  - Teva Investigational Site 54245, Jindřichův Hradec
  - Teva Investigational Site 54244, Teplice
  - Teva Investigational Site 54243, Varnsdorf
- Germany (9):
  - Teva Investigational Site 32881, Ahrensburg
  - Teva Investigational Site 32880, Bendorf
  - Teva Investigational Site 32884, Berlin
  - Teva Investigational Site 32879, Frankfurt
  - Teva Investigational Site 32883, Leipzig
  - Teva Investigational Site 32876, Leipzig
  - Teva Investigational Site 32877, Magdeburg
  - Teva Investigational Site 32878, Mainz A. Rhein
  - Teva Investigational Site 32882, Rheine
- Israel (3):
  - Teva Investigational Site 80207, Be’er Ya‘aqov
  - Teva Investigational Site 80206, Haifa
  - Teva Investigational Site 80208, Jerusalem
- Mexico (5):
  - Teva Investigational Site 21133, Chihuahua City
  - Teva Investigational Site 21134, Mexico City
  - Teva Investigational Site 21137, Morelia
  - Teva Investigational Site 21136, Tlalnepantla
  - Teva Investigational Site 21135, Zapopan
- Poland (5):
  - Teva Investigational Site 53578, Gdansk
  - Teva Investigational Site 53575, Lodz
  - Teva Investigational Site 53576, Lodz
  - Teva Investigational Site 53574, Tarnów
  - Teva Investigational Site 53577, Wroclaw
- Romania (3):
  - Teva Investigational Site 52148, Craiova
  - Teva Investigational Site 52147, Oradea
  - Teva Investigational Site 52145, Timișoara
- Slovakia (3):
  - Teva Investigational Site 62102, Košice
  - Teva Investigational Site 62103, Martin
  - Teva Investigational Site 62101, Spišská Nová Ves
- Turkey (Türkiye) (4):
  - Teva Investigational Site 82089, Adana
  - Teva Investigational Site 82088, Kocaeli
  - Teva Investigational Site 82085, Kırıkkale
  - Teva Investigational Site 82087, Mersin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be assessed for scientific merit, product approval status, and conflicts of interest. If the request is approved, patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.